CLINICAL TRIAL: NCT03413774
Title: Unexplained Early Miscarriage : Role and Prevalence of Lower Genital Tract Infections in Rural Area in Egypt
Brief Title: Unexplained Early Miscarriage : Role and Prevalence of Lower Genital Tract Infections
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Other Study IDs: 24
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: First Trimester Abortion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abortion group: 910 women attended Fayoum University hospital outpatient gynecology clinic with recent first trimesteric spontaneous miscarriage
  Interventions: Procedure: vaginal swab
- Control group: 940 women attended Fayoum University hospitalpresented for any other gynecological complaint
  Interventions: Procedure: vaginal swab

INTERVENTIONS:
Procedure: vaginal swab — high vaginal and Endocrvical swabs for bacterial, protozoal and chlamydial infection- examined by PCR
  Other Names: high vaginal swab

SUMMARY:
The study group included 910 women who attended Fayoum university hospital gynecology outpatient clinic for postabortive evaluation. The control group included 940 women attended outpatient clinic for any other procedure or complaint

DETAILED DESCRIPTION:
The study group included 910 women who attended Fayoum university hospital gynecology outpatient clinic for postabortive evaluation. The control group included 940 women attended outpatient clinic for any other procedure or complaint all patients were screened by serum samples to detect IgM / IgG to Chlamydia trachomatis (DRG Chlamydia Trachomatis IgM / IgG Enzyme immunoassay) and by high vaginal and Endocrvical swabs for bacterial, protozoal and chlamydial infection- examined by PCR- (from +ve samples to chlamydial IgM / IgG).

ELIGIBILITY:
Inclusion Criteria:

* The Study group included Women with recent unexplained early miscarriage (pregnancy duration 12 weeks or less and miscarriage within 4 weeks)
* The control group included Women with any other gynecological complaint or in need of family planning

Exclusion Criteria:

* Miscarriage of Pregnancy duration more than 12 ws Documented causes of miscarriage as fetal or uterine anomalies, antiphospholipid syndrome, endocrine factors….etc
* Recent antibiotic, antifungal or antiprotozoal treatment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: * The Study group included Women with recent unexplained early miscarriage (pregnancy duration 12 weeks or less and miscarriage within 4 weeks)
  * The control group included Women with any other gynecological complaint or in need of family planning
Sampling Method: Non-Probability Sample
Enrollment: 1850 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
prevalence of lower genital tract infection | At time of examination
  candida, bacterial vaginosis , trichomonas , mycoplasmal or chlamydial infection

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No